CLINICAL TRIAL: NCT06095375
Title: Regorafenib in Combination With Temozolomide With or Without Radiotherapy in Patients With Newly Diagnosed MGMT-Methylated, IDH Wild-type Glioblastoma. A Phase I Dose-finding Study
Brief Title: Regorafenib With Temozolomide With or Without RT in MGMT-Methylated, IDH Wild-type GBM Patients
Acronym: REGOMA-2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Collaborators: Bayer S.p.A (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IOV-GB-1-2021-REGOMA2; 2021-001604-15 (EudraCT Number)
Record Dates: First submitted 2023-03-10; First posted 2023-10-23 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma, IDH-wildtype; MGMT-Methylated Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — regorafenib; Temozolomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A (Adjuvant/Maintenance Phase) (Experimental)
  Interventions: Drug: Regorafenib; Drug: Temozolomide
- Cohort B (Concomitant Phase) (Experimental)
  Interventions: Drug: Regorafenib; Drug: Temozolomide

INTERVENTIONS:
Drug: Regorafenib — Cohort A (Adjuvant/Maintenance Phase). The Adjuvant (Maintenance) Therapy dose escalation will explore three dose levels of regorafenib (e.g., 80 mg, 120 mg and 160 mg; level-1: regorafenib 40 mg will be evaluated in case of DLT during regorafenib 80 mg) administered in combination with adjuvant TMZ to evaluate the initial toxicity of regorafenib and TMZ Cohort B (Concomitant Phase) Therapy dose escalation will explore three dose levels of regorafenib (e.g., 80 mg, 120 mg and 160 mg; level -1: regorafenib 40 mg will be evaluated in case of DLT during regorafenib 80 mg) administered in combination with TMZ and RT.
Drug: Temozolomide — Following a "3+3" design, in cohort A three patients will be administered temozolomide 150-200 mg/m2 for 5 consecutive days every 28 days until 6-12 cycles and regorafenib daily for 21 days, with a 1-week washout period at dose of 80 mg (level 1), 120 mg (level 2), or 160 mg (level 3) (regorafenib 40 mg- level -1). As a general rule, one cycle will last 28 days (day 1-28); however, in the event of treatment prolongation, the cycle period will be extended.
  In cohort B,During concomitant therapy phase: temozolomide 75 mg/m2/die for 42 (max 49 days) consecutive days (concomitant with radiation therapy).

SUMMARY:
This study will evaluate the addition of regorafenib to standard of care treatment with TMZ as adjuvant therapy, and in combination with TMZ+RT as concomitant therapy.

The standard of care for newly diagnosed GBM (ndGBM) includes surgical resection to the extent that is safely feasible, followed by RT plus concomitant TMZ chemotherapy, and up to 6 months of adjuvant TMZ.

The dose escalation will be explored following a "3+3" design, escalating oral doses of regorafenib in combination with adjuvant (maintenance) TMZ (cohort A) to estimate the MTD of regorafenib as adjuvant (maintenance) therapy. After finding the MTD in the Adjuvant Therapy dose escalation, the Concomitant Therapy (cohort B) dose escalation will start, exploring escalating oral doses of regorafenib in combination with concomitant TMZ+RT, to estimate the MTD of regorafenib as concomitant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of ≥ 18 years of age at the time of signing the informed consent form (ICF).
* Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted
* Patients capable of taking oral medication
* Subject is willing and able to adhere to the study visit schedule and other protocol requirements.
* Histologically confirmed Grade IV GBM/gliosarcoma (WHO criteria; non-IDH R132Hmutant by immunohistochemistry [IHC] or, sequencing for IDH1 and 2 in case of patients >55 years) established following either a radical or partial surgical resection. This includes treatment naïve (chemotherapy and RT) patients with prior histologically diagnosis of lower-grade astrocytoma that has been upgraded to a histologically verified glioblastoma after a subsequent definitive surgery.

NOTE: Patients with known isocitrate dehydrogenase (IDH) 1 and 2 are to be excluded.

* Methylated MGMT according to local laboratory (in case of pyrosequencing, methylation >10%)
* Subject must have recovered from the effects of surgery, including post-operative infections or complications. Toxicities resulting from surgery must have resolved to NCI CTCAE (v5.0) Grade ≤ 1 prior to starting regorafenib treatment (with the exception of Grade 2 alopecia).
* For Concomitant Therapy Cohort: Prior tumor resection up to 7 weeks prior to the first dose of regorafenib.
* For Adjuvant Therapy Cohort: Subject must have recently completed standard course of radiotherapy with TMZ chemotherapy, and then have an MRI documenting stable disease prior to the first dose of regorafenib (In case of "pseudoprogression" the patient will not be eligible)
* For Adjuvant Therapy:

  1. All AEs resulting from prior RT+TMZ chemotherapy must have resolved to NCI CTCAE (v5.0) Grade 1 (except for laboratory parameters outlined below).
  2. Subject must have not experienced significant toxicity to prior RT+TMZ (i.e., Grade 4 hematological toxicity)
* Subjects must have life expectancy of at least 6 months
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 to 1 (or KPS 70)
* Corticosteroid use of dexamethasone 4 mg or less per day within 7 days before starting regorafenib.
* Subject must have the following laboratory values at screening within 7 days before starting regorafenib:

  1. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L without growth factor support for 7 days (14 days if subject received pegfilgrastim).
  2. Hemoglobin (Hgb) ≥10 g/dL
  3. Platelet count (plt) ≥100x 109/L
  4. Serum potassium concentration within normal range, or correctable with supplements
  5. Serum glutamic oxaloacetic transaminase (SGOT)/aspartate aminotransferase (AST) and serum glutamate pyruvic transaminase (SGPT)/alanine aminotransferase (ALT) ≤ 3.0 x Upper Limit of Normal (ULN).
  6. Serum total bilirubin ≤ 1.5 x ULN
  7. Serum creatinine ≤ 1.5 x ULN or measured glomerular filtration rate (GFR) ≥ 50 mL/min/1.73 m2 using an exogenous filtration marker such as iohexol, inulin, 51Cr EDTA or 1125 iothalamate, or creatinine clearance of ≥ 50 mL/min using Cockroft-Gault equation.
  8. Serum albumin > 3.5 g/dL
  9. PT (or INR) and APTT within normal range
* For women who are not postmenopausal (i.e., < 2 years after last menstruation) or surgically sterile (absence of ovaries and/or uterus) and who are sexually active: agreement to use an adequate method of contraception (oral contraceptives, intrauterine contraceptive device, or barrier method of contraception in conjunction with spermicidal jelly) during the Treatment period and for at least 6 months after the last dose of study drug.
* For male patients who are partners of premenopausal women: agreement to use a barrier method of contraception during the Treatment period and for at least 6 months after the last dose of study drug.

Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are eligible to participate.

Exclusion Criteria:

* Received any prior treatment for glioma including:

  1. Prior prolifeprospan 20 with carmustine wafer.
  2. Prior intracerebral agent.
  3. Prior radiation treatment for GBM or lower-grade glioma.
  4. Prior chemotherapy or immunotherapy for GBM or lower-grade glioma.
  5. NOTE: 5-aminolevulinic acid-mediated photodynamic therapy and Flourcrescein administered prior to surgery to aid in optimal surgical resection is not considered a chemotherapy agent.
* Patients who performed biopsy as surgical approach of glioblastoma.
* Patients who are taking strong cytochrome P (CYP) CYP3A4 inhibitors (eg, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, telithromycin, voriconazole) or strong CYP3A4 inducers (eg, carbamazepine, phenobarbital, phenytoin, rifampin, St. John's Wort).
* Patients who are receiving additional, concurrent, active therapy for GBM outside of the trial.
* Disease located outside of the brain (e.g. brainstem and leptomeningeal disease).
* Candidate for urgent palliative intervention for primary disease (e.g., impending herniation) as judged by the Investigator
* History of allergy or hypersensitivity to any of the study treatments or any of their excipients.
* In the presence of therapeutic intent to anticoagulate the patient: INR or PT and aPTT not within therapeutic limits (according to the medical standard in the institution). NOTE: Per American Society of Clinical Oncology (ASCO) guidelines, use of low-molecular-weight heparin (LMWH) should be the preferred approach.
* Unable or unwilling to undergo brain MRI scans with intravenous (IV) gadolinium.

History of another malignancy in the previous 3 years, with a disease-free interval of< 3 years. Patients with prior history of in situ cancer or basal or squamous cell skin cancer are eligible.

* Serious, non-healing wound, ulcer, bone fracture, or abscess.
* Any cerebrovascular accident (including transient ischemic attacks) within the last 6 months prior to initiation of study treatment.
* Have an ongoing infection with severity of Grade 2 or above (CTCAE 5.0)
* Any hemorrhage or bleeding event that is ≥ Grade 3 based on the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Event (CTCAE), Grade 2 intracranial hemorrhage, or persistent thrombotic/embolic event within 4 weeks prior to the start of study medication.
* Uncontrolled or severe cardiac disease (e.g., history of unstable angina, myocardial infarction, coronary stenting, or bypass surgery within the last 6 months prior to initiation of study treatment), symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia (including atrial flutter/fibrillation), requirement for inotropic support or use of devices for cardiac conditions (e.g., pacemakers/defibrillators), or hypertension (participants with systolic blood pressure[BP] of > 160 mmHg or diastolic BP of > 100 mmHg despite optimal medical management are to be excluded).
* History of interstitial lung disease, history of slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis, or symptomatic pleural effusion.
* Active, known, or suspected auto-immune disease, including systemic lupus erythematosus, Hashimotos thyroiditis, scleroderma, polyarteritis nodosa, or auto-immune hepatitis.
* Known history of hepatitis B, human immunodeficiency virus (HIV), or active hepatitis C infection requiring treatment with antiviral therapy. Note: HIV testing is not required in the absence of clinical suspicion.
* History of bleeding diathesis (irrespective of severity).
* Uncontrolled intercurrent illness including (e.g., symptomatic ascites), but not limited to ongoing or active infection.
* Persistent ≥ Grade 3 Lipase (> 2.0 - 5.0 x upper limit of normal [ULN] with signs or symptoms; > 5.0 x ULN and asymptomatic).
* Persistent proteinuria> 3.5 g/24 hours measured by urine protein creatinine ratio from a random urine sample (≥ Grade 3, CTCAE 5.0)
* Have any malabsorbition condition.
* Any condition that could make the subject noncompliant with the study procedures and/or study requirements, as judged by the Investigator (for example: cognitive impairment, psychiatric illness, etc).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2024-10-09 (Actual); Study Completion 2025-12-22 (Actual)

PRIMARY OUTCOMES:
Number of patients with a Dose Limiting Toxicity (DLT) | During dose escalation, the DLT evaluation period will be two cycles from Day -1 of Cycle 1 of adjuvant phase (cohort A) or from Day 1 to last day of the concomitant RT phase (Cohort B). (each cycle is 28 days)
Number of patients with ≥1 adverse event (AE) using the NCI CTCAE v5.0 | evaluation period will be two cycles from Day -1 of Cycle 1 of adjuvant phase (cohort A) or from Day 1 to last day of the concomitant RT phase (Cohort B). (each cycle is 28 days)
  * Grade 3 diarrhea, nausea, vomiting, and loss of appetite if lasting for ≥ 7 consecutive days;
  * Grade 3 electrolyte imbalance if lasting for ≥ 7 consecutive days;
  * Grade 3 dermal toxicity if lasting for ≥ 7 consecutive days;
  * Grade 3 fatigue for ≥ 7 consecutive days;
  * Grade 4 T-Bil, AST (GOT) and/or ALT (GPT) elevations,
Number of patients discontinuing study treatment due to an AE | evaluation period will be two cycles from Day -1 of Cycle 1 of adjuvant phase (cohort A) or from Day 1 to last day of the concomitant RT phase (Cohort B). (each cycle is 28 days)
  Number of patients discontinuing study treatment due to an AE

SECONDARY OUTCOMES:
Pharmacokinetics parameters - AUC | evaluation period will be two cycles from Day -1 of Cycle 1 of adjuvant phase (cohort A) or from Day 1 to last day of the concomitant RT phase (Cohort B). (each cycle is 28 days)
  area under the plasma concentration versus time curve
Best response to treatment according to RANO criteria | from date of randomization until the date of first occurrence of disease progression or death, whichever come first,assessed up to 32 months
  Tumor response according to RANO criteria
Progression-free survival | from the start of radiotherapy until the date of first occurrence of disease progression or death whichever come first,assessed up to 32 months
  Survival time without tumor progression
EORTC QLQ-C30 | from the start of radiotherapy until the date of first occurrence of disease progression or death whichever come first,assessed up to 32 months
  Survey with evaluations at screening, concurrently to brain MRI assessment and at the end of treatment
Pharmacokinetics parameters - Tmax | evaluation period will be two cycles from Day -1 of Cycle 1 of adjuvant phase (cohort A) or from Day 1 to last day of the concomitant RT phase (Cohort B). (each cycle is 28 days)
  Time to peak drug concentration
Pharmacokinetics parameters - Cmax | evaluation period will be two cycles from Day -1 of Cycle 1 of adjuvant phase (cohort A) or from Day 1 to last day of the concomitant RT phase (Cohort B). (each cycle is 28 days)
  Peak plasma concentration
Overall survival | from the start of radiotherapy until death ,assessed up to 32 months
Brain module BN20 | from the start of radiotherapy until the date of first occurrence of disease progression or death whichever come first,assessed up to 32 months
  Survey with evaluations at screening, concurrently to brain MRI assessment and at the end of treatment

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Istituto Oncologico Veneto IRCCS, Padua
  - Humanitas Research Hospital, Rozzano